CLINICAL TRIAL: NCT01123226
Title: Relative Effectiveness of Trigger Point Therapy Compared to Spinal Manipulation in Correcting a Thoracic Spinal Manipulable Lesion in Subjects With Mechanical Thoracic Back Pain: a Randomised Trial
Brief Title: Trigger Point Therapy Versus Manipulation Correcting Thoracic Manipulable Lesion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anglo-European College of Chiropractic (Other)
Responsible Party: Hugh Gemmell Principal Lecturer, Anglo-European College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AECC05052010
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Spinal Manipulable Lesion; Somatic Dysfunction
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diversified HVLA spinal manipulation (Experimental)
  Interventions: Procedure: spinal manipulation
- Trigger point pressure release (Active Comparator)
  Interventions: Procedure: trigger point therapy

INTERVENTIONS:
Procedure: spinal manipulation — A maximum of two high velocity low amplitude spinal manipulations to one dysfunctional spine joint
  Arms: Diversified HVLA spinal manipulation
Procedure: trigger point therapy — The thumb will apply firm pressure to a trigger point in the paravertebral multifidus and rotatores muscles associated with the spine joint dysfunction using the barrier approach. This will be held until the barrier releases and this will continue until the trigger point is inactivated or 3 minutes has passed.
  Arms: Trigger point pressure release

SUMMARY:
There will be no difference between trigger point therapy and spinal manipulation in correcting a spine joint dysfunction in the back

ELIGIBILITY:
Inclusion Criteria:

* mechanical thoracic back pain
* age 18-64
* presence of at least one spinal manipulable lesion
* presence of a trigger point associated with the spinal manipulable lesion
* able to lie prone on a treatment table for 15 minutes

Exclusion Criteria:

* absolute contraindications to spinal manipulation
* specific thoracic back pain
* bleeding diathesis, use of anticoagulants, long-term corticosteroid use
* involved in litigation for thoracic back pain
* inability to read or write English fluently
* treatment with manipulation or myofascial therapy within past three days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Correction of spinal manipulable lesion | Immediate effect of one treatment
  Dichotomous data either lesion is corrected or not.

SECONDARY OUTCOMES:
Change in pressure pain threshold over the involved spinous process | Immediate effect of one treatment
  The point at which sensation changes from that of pressure to pain is measured in Kg/cm2

CONTACTS AND LOCATIONS:
Locations (1):
- Anglo-European College of Chiropractic, Bournemouth, Dorset, United Kingdom